CLINICAL TRIAL: NCT06632353
Title: Biomarkers in Dermal Interstitial Fluid for Early Diagnosis and Follow-up of Cardiovascular Diseases
Acronym: BIO-ISF-CVD
Status: Active, not recruiting | Type: Observational
Sponsor: Ascilion AB (Industry)
Responsible Party: Sponsor
Other Study IDs: CIV-23-08-043912
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — dISF sample, plasma sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Cardiovascular diseases
- Group 2: Reference

SUMMARY:
Sampling of dISF and blood plasma for qualitative measurements.

DETAILED DESCRIPTION:
Sampling of dISF will be performed to investigate biomarkers in dISF for early diagnosis and follow-up of cardiovascular diseases.

ELIGIBILITY:
Inclusion criteria:

Group 1: Chronic heart failure with stable therapy. NYHA classification II, III and IV. Age > 60 years. Group 2: Age 18-40 years.

Exclusion criteria:

* Participating in another clinical investigation which may affect the study outcome according to clinical judgement.
* Previous use of sampling system used.
* Pregnancy or lactating.
* Any disease or condition that may be affected.
* Individuals who lack the ability to fully consent to participate in the study.
* Severe skin injury.
* Tattoo or piercing close to sampling area.
* Group 1: All forms of emergency care.
* Group 1: Non-stable therapy.
* Group 1: Sepsis.
* Group 1: BMI > 30kg/m2.
* Group 1: Age > 84 years.
* Group 2: Known heart or vascular disease.
* Group 2: Diabetes.
* Group 2: Kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and subjects recruited at hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of dISF biomarker | Day 1
  Presence or not

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyd Hospital, Danderyd, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Will probably be published